CLINICAL TRIAL: NCT01912378
Title: Phase 1 Study of Intranasal Oxytocin on Parents' Behavioral and Physiological Responses to Children With Autism
Brief Title: Triadic Interactions of Families With Autism and Oxytocin
Acronym: TAO
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to launch the study due to lack of participation with Autism Clinic
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TAO
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Autism Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin Nasal Spray (Experimental): 40 IUs of Oxytocin nasal spray will be administered to both parents at one time during the lab visit.
  Interventions: Drug: Oxytocin
- Placebo nasal spray (Placebo Comparator): 40 IUs of Placebo nasal spray will be administered to both parents at one time during the lab visit.
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Novartis
  Arms: Oxytocin Nasal Spray
Drug: Placebo nasal spray
  Arms: Placebo nasal spray

SUMMARY:
The study will investigate the effects of an intranasal administration of oxytocin (OT) to parents of children with autism spectrum disorders (ASD) on the quality of mother-father-child interactions. Physiological and behavioral measures of parent-child triadic interaction quality will be assessed.

H1: Parents who receive OT will demonstrate greater parental engagement and nonverbal prosocial behaviors compared to parents who receive placebo.

H2: Children with ASD whose parents receive OT will have increased nonverbal prosocial behaviors during the discussion and play tasks compared to children whose parents' receive placebo.

H3: Parents who receive OT will demonstrate increased behavioral and physiological synchrony with their child during the discussion and play tasks compared to parents who receive placebo and their child.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a continuum of neurodevelopmental disorders associated with significant communication, social, and behavioral deficits including impairments in verbal and nonverbal communication and excessive attachments to routine. These deficits can impede parent-child bonding, increase parental stress, and lead to dysfunctional parent-child interactions. While there has been progress into understanding the neurobiology and neuropsychology of schizophrenia and autism spectrum disorder, treatment options remain inadequate. Psychosocial interventions such as family therapy aimed at promoting affection, praise, and communication reduce oppositional behavior, but are time consuming and costly. A safe and cost-effective pharmacological intervention given to non-affected family members could augment current psychosocial therapies, improve the functioning of the family, and favorably influence the course of the illness in the affected child.

Oxytocin (OT) is a neuropeptide associated with parenting and social perception in mammals. Exogenous OT can be safely administered intranasally in humans, enters the brain in high concentrations, increases positive interpersonal and parenting interactions, promotes cooperation and trust, and reduces stress-induced physiological responses. Due to OT's involvement in processes associated with parent-child interactions (e.g. bonding), we hypothesize that the OT system represents a highly promising focus of research into the biological underpinnings of family functioning, as well as a promising target for biological interventions aimed at improving communication between parents and their children with ASD and reducing unhealthy interactions. We will test these hypotheses by exploring the effects of exogenously administered OT to caregivers on parent-child interactions and physiology during a laboratory-based parent-child interaction task. If successful, this would represent the first demonstration of a neurobiological factor in the family functioning of persons with ASD, and would represent the first biological intervention applied to family members of persons with ASD, rather than to the individual with ASD.

The purpose of the current study is twofold: 2) To determine whether administration of the affiliative neuropeptide oxytocin to the parent positively influences parent-child interactions of patients with autism spectrum disorders, and 2) to explore the mechanisms by which parental behavior affects children's behavior, feelings, and physiology.

Participants will be 40 triads consisting of mother, father, and child with ASD and 40 triads of mother, father, and typically developing (TD) children. Families will come to our lab at UCSF's Parnassus campus for one 2-hour visit. Parent dyads will be randomly assigned to receive either OT or placebo immediately before the triad engages in triadic discussion and play tasks. We will monitor mothers', fathers', and children's physiological and behavioral responses during these tasks. In summary, this is a randomized 2 (diagnosis) x 2 (spray) between-subjects study of triadic physiology and behavior in children with ASD or TD in which both mothers and fathers are given either OT or placebo.

ELIGIBILITY:
Inclusion Criteria:

For parents of patients with ASD and TD controls:

* Age between 25 and 60 years old
* Live with child
* Read and communicate in English

For patient with ASD:

* Age between 7 and 12 years old
* Lives with parents
* Has diagnosis of autism spectrum disorder, pervasive developmental disorder, or pervasive developmental disorder-not otherwise specified(PDD-NOS)
* Communicates in English
* Has IQ at or above 75

For TD controls:

* Age between 7 and 12 years
* Lives with parents

Exclusion Criteria:

For parents of patients with ASD and TD controls:

* Female parents who state they are pregnant or have a positive pregnancy test
* Severe psychiatric, neurologic or medical illness
* Severe nasal pathology, atrophic rhinitis, recurrent nose bleeds, or history of cranial-surgical procedures (hypophysectomy)
* History of severe psychiatric diagnosis including schizophrenia, bipolar, and autism
* Divorce or separation
* Hypertension, pacemaker, cardiovascular medications

For patients with ASD:

* IQ lower than 75

For TD controls:

* Current psychiatric illness or developmental disability
* Current psychiatric medication

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Parental social behavior | 37 minutes into lab visit
  Social engagement behaviors, including postural orientation, high gaze, quality and quantity of language directed toward child, facial expressions of affect.

SECONDARY OUTCOMES:
Child and Parent Physiological Synchrony | 32 minutes into lab visit
  Sympathetic, parasympathetic, and neuroendocrine responses of both parents and child.
Child social behavior | 37 minutes into lab visit
  Social engagement behaviors, including postural orientation, high gaze, quality and quantity of language directed toward parent, facial expressions of affect.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Mendes, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Abidin, R. R. (1995). Parenting Stress Index, Third Edition. Professional Manual. Odessa, FL.: Psychological Assessment Resources, Inc.
- [Background] Achenbach, T. (2001). Manual for the Child Behavior Checklist/4-18. Burlington, VT: University of Vermont.
- [Background] Aron, A., Aron, E. N., & Smollan, D. (1992). Inclusion of other in the self scale and the structure of interpersonal closeness. Journal of Personality and Social Psychology, 63, 596-612.
- [Background] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Background] Buchheim A, Heinrichs M, George C, Pokorny D, Koops E, Henningsen P, O'Connor MF, Gundel H. Oxytocin enhances the experience of attachment security. Psychoneuroendocrinology. 2009 Oct;34(9):1417-22. doi: 10.1016/j.psyneuen.2009.04.002. Epub 2009 May 19. PMID 19457618
- [Background] Busby, D. M., Christensen, C., Crane, D. R., & Larson, J. H. (1995). A revision of the Dyadic Adjustment Scale for use with distressed and nondistressed couples: Construct hierarchy and multidimensional scales. Journal of Marital and Family Therapy, 21, 289-308.
- [Background] Ditzen B, Schaer M, Gabriel B, Bodenmann G, Ehlert U, Heinrichs M. Intranasal oxytocin increases positive communication and reduces cortisol levels during couple conflict. Biol Psychiatry. 2009 May 1;65(9):728-31. doi: 10.1016/j.biopsych.2008.10.011. Epub 2008 Nov 22. PMID 19027101
- [Background] Feldman R, Gordon I, Zagoory-Sharon O. The cross-generation transmission of oxytocin in humans. Horm Behav. 2010 Sep;58(4):669-76. doi: 10.1016/j.yhbeh.2010.06.005. Epub 2010 Jun 15. PMID 20558167
- [Background] Gordon I, Zagoory-Sharon O, Schneiderman I, Leckman JF, Weller A, Feldman R. Oxytocin and cortisol in romantically unattached young adults: associations with bonding and psychological distress. Psychophysiology. 2008 May;45(3):349-52. doi: 10.1111/j.1469-8986.2008.00649.x. Epub 2008 Feb 4. PMID 18266803
- [Background] Gordon I, Zagoory-Sharon O, Leckman JF, Feldman R. Oxytocin and the development of parenting in humans. Biol Psychiatry. 2010 Aug 15;68(4):377-82. doi: 10.1016/j.biopsych.2010.02.005. Epub 2010 Mar 31. PMID 20359699
- [Background] Gouin JP, Carter CS, Pournajafi-Nazarloo H, Glaser R, Malarkey WB, Loving TJ, Stowell J, Kiecolt-Glaser JK. Marital behavior, oxytocin, vasopressin, and wound healing. Psychoneuroendocrinology. 2010 Aug;35(7):1082-90. doi: 10.1016/j.psyneuen.2010.01.009. Epub 2010 Feb 9. PMID 20144509
- [Background] Grewen KM, Girdler SS, Amico J, Light KC. Effects of partner support on resting oxytocin, cortisol, norepinephrine, and blood pressure before and after warm partner contact. Psychosom Med. 2005 Jul-Aug;67(4):531-8. doi: 10.1097/01.psy.0000170341.88395.47. PMID 16046364
- [Background] Heinrichs M, Baumgartner T, Kirschbaum C, Ehlert U. Social support and oxytocin interact to suppress cortisol and subjective responses to psychosocial stress. Biol Psychiatry. 2003 Dec 15;54(12):1389-98. doi: 10.1016/s0006-3223(03)00465-7. PMID 14675803
- [Background] Kerns KA, Aspelmeier JE, Gentzler AL, Grabill CM. Parent-child attachment and monitoring in middle childhood. J Fam Psychol. 2001 Mar;15(1):69-81. doi: 10.1037//0893-3200.15.1.69. PMID 11322086
- [Background] Light KC, Grewen KM, Amico JA. More frequent partner hugs and higher oxytocin levels are linked to lower blood pressure and heart rate in premenopausal women. Biol Psychol. 2005 Apr;69(1):5-21. doi: 10.1016/j.biopsycho.2004.11.002. Epub 2004 Dec 29. PMID 15740822
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- [Background] Naber F, van Ijzendoorn MH, Deschamps P, van Engeland H, Bakermans-Kranenburg MJ. Intranasal oxytocin increases fathers' observed responsiveness during play with their children: a double-blind within-subject experiment. Psychoneuroendocrinology. 2010 Nov;35(10):1583-6. doi: 10.1016/j.psyneuen.2010.04.007. Epub 2010 May 8. PMID 20457491
- [Background] Radloff, L. S. (1977). The CES-D Scale. A self-report depression scale for research in the general population. Applied Psychological Measurement, 1, 385-401.
- [Background] Theodoridou A, Rowe AC, Penton-Voak IS, Rogers PJ. Oxytocin and social perception: oxytocin increases perceived facial trustworthiness and attractiveness. Horm Behav. 2009 Jun;56(1):128-32. doi: 10.1016/j.yhbeh.2009.03.019. Epub 2009 Apr 1. PMID 19344725
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wei M, Russell DW, Mallinckrodt B, Vogel DL. The Experiences in Close Relationship Scale (ECR)-short form: reliability, validity, and factor structure. J Pers Assess. 2007 Apr;88(2):187-204. doi: 10.1080/00223890701268041. PMID 17437384